CLINICAL TRIAL: NCT05368181
Title: The MAGIC Algorithm Probability Guided Preemption of Steroid-refractory Graft-versus-host Disease With Methylprednisolone
Brief Title: MAP-guided Preemptive Therapy of aGvHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Primary investigator, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HXMAP 1.0
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: GVHD,Acute; Stem Cell Transplant Complications
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: methylprednisolone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention group (Experimental): Methylprednisolone starts with the dose of 2 mg/kg for 5 days. If no signs of aGvHD, the dose of methylprednisolone is gradually taper with the following 16 days.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone starts with the dose of 2 mg/kg for 5 days. If no signs of aGvHD, the dose of methylprednisolone is gradually taper with the following 16 days.

SUMMARY:
Acute graft versus host disease (aGvHD) is a severe and potentially fatal complication of allogeneic hematopoietic stem cell transplantation (HCT). The Mount Sinai Acute GVHD International Consortium (MAGIC) algorithm probability (MAP) identifies patients who are at high risk for severe aGvHD as early as 7 days after HCT based on 2 serum biomarkers, suppressor of tumorigenesis 2 (ST2) and regenerating islet-derived 3α (Reg3α). Patients who consent to this study will have their blood tested weekly up to four times within the first month post HCT to determine if they are at high risk for severe GVHD based on MAP. Patients who are at high risk at any of these four tests will be treated with methylprednisolone to see if it prevents the development of severe aGvHD. Methylprednisolone starts with the dose of 2 mg/kg for 5 days. If no signs of aGvHD, the dose of methylprednisolone is gradually tapered within the following 16 days. Patients will be followed for the development of severe aGvHD for up to 3 months from the HCT and will continue to be followed at routine clinic visits for up to one year after HCT.

ELIGIBILITY:
Inclusion Criteria:

* Any donor type (e.g., related, unrelated, haplo) or stem cell source (bone marrow, peripheral blood, cord blood).
* Any conditioning regimen (non-myeloablative, myeloablative, or reduced intensity) is acceptable.
* GVHD prophylaxis must include a calcineurin inhibitor combined with post transplant cyclophosphamide.
* The use of serotherapy to prevent GVHD (e.g., antithymocyte globulin) prior to day 3 post-HCT is permitted
* Direct bilirubin must be <2 mg/dL unless the elevation is known to be due to Gilbert syndrome within 3 days prior to enrollment.
* ALT/SGPT and AST/SGOT must be <5 x the upper limit of the normal range within 3 days prior to enrollment.
* Signed and dated written informed consent obtained from patient or legal representative.

Exclusion Criteria:

* Patients who develop acute GVHD prior to start of study drug
* Patients at very high risk for relapse post HCT as defined by very high disease risk index
* Patients participating in a clinical trial where prevention of GVHD is the primary endpoint
* Uncontrolled active infection (i.e., progressive symptoms related to infection despite treatment or persistently positive microbiological cultures despite treatment or any other evidence of severe sepsis)
* Patients who are pregnant
* Patients on dialysis within 7 days of enrollment
* Patients requiring ventilator support or oxygen supplementation exceeding 40% FiO2 within 14 days of enrollment.
* Patients receiving investigational agent within 30 days of enrollment. However, the Principal Investigator (PI) may approve prior use of an investigational agent if the agent is not expected to interfere with the safety or the efficacy of methylprednisolone.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of High Risk Patients Who Develop Grade III or IV aGvHD | Day 100 post HCT
  Number of High Risk Patients Who Develop Grade III or IV aGvHD by day 100 post HCT

SECONDARY OUTCOMES:
Number of Participants Alive at 6 Months and 1 Year | 6 months and 1 year
  Overall survival - The number of that patients are still alive from the start of treatment at 6 months and 1 year
Number of Participants With Non-relapse Mortality (NRM) | 6 months and 1 year
  Number of participants with NRM - deaths which could not be attributed to disease relapse or progression. Non-relapse mortality defined as death without prior relapse.
Number of Participants With Relapse | 1 year
  Number of participants with relapse at one year. Relapse defined as recurrence of disease that required transplant.
Number of Participants With Clinically Relevant GVHD States Grade II-IV GVHD | 100 days
  Number of participants with clinically relevant GVHD states grade II-IV GVHD requiring systemic treatment.
Number of Participants With Chronic GVHD Requiring Systemic Steroid Treatment | 1 year
  Number of participants with chronic GVHD requiring systemic steroid treatment. Chronic GVHD Requiring Systemic Steroid Treatment: defined as the development of symptoms of chronic GVHD according to NIH Consensus Criteria that require treatment with oral or intravenous corticosteroids.
Number of Participants With Serious Infections | 1 year
  Number of participants with serious infections (defined as grade 3 by the Blood and Marrow Transplant Clinical Trials Network). Serious Infection: Defined as bacterial, fungal, viral or parasitic infections that required oral or intravenous treatments such as antibiotics.
Overall survival | 1 year
  Overall survival of this group of patients at the end of 1 year
GvHD free and relapse free survival | 1 year
  Survival of patients without grade 3 or 4 aGvHD or disseminated cGvHD or relapse of disease at end of 1 year post HCT

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No